CLINICAL TRIAL: NCT04365777
Title: EEG Characteristics of Different Sedation Depths in Patients With Supratentorial Glioma in Frontal Lobe
Brief Title: EEG Characteristics of Different Sedation Depths in Neurosurgery Patients
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, professor, Beijing Tiantan Hospital
Other Study IDs: ChiECRCT20200002
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Electroencephalography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Awake State: OAA/S=5
  Interventions: Other: OAA/S=5
- Sedation State: OAA/S=3
  Interventions: Other: OAA/S=3
- Unconsciousness State: OAA/S=1
  Interventions: Other: OAA/S=1

INTERVENTIONS:
Other: OAA/S=5 — Prior to anesthesia induciton, EEG signatures will be recorded at Observer's Assessment of Alertness/Sedation (OAA/S) score of 5 (awake, eye-close state) for few minutes.
  Groups: Awake State
Other: OAA/S=3 — Given sedative anesthetics (propofol, midazolam or dexmetomidine), EEG signatures will be recorded after reaching steady state of OAA/S=3 (responds only after name called loudly and/or repeatedly) for few minutes.
  Groups: Sedation State
Other: OAA/S=1 — Increasing drug concentration, EEG signatures will be recorded after reaching steady state of OAA/S=1 (does not respond to noxious stimuli) for few minutes.
  Groups: Unconsciousness State

SUMMARY:
Gliomas are the most common primary intracranial malignancy, and behavioral experiments in patients with supratentorial gliomas under sedation have shown potential neurological abnormalities; however, these behavioral experiments are susceptible to external influences. Therefore, more objective evidence is needed to support and extend the existing conclusions. The purpose of this study is to compare the EEG signatures (such as the EEG signal power) at various levels of anesthetics induced sedation in patients with supratentorial glioma in frontal lobe and in patients without intracranial-occupying lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with supratentorial glioma in right frontal lobe, and patients requiring general anesthesia without intracranial-occupying lesion;
2. Aged 18-60 years;
3. ASA I to II;
4. All those who sign the informed consent form.

Exclusion Criteria:

1. Obese patients, BMI>30kg/m2;
2. Patients with Mallampati class III to IV airway anatomy;
3. Combined with other neurological or psychiatric diseases;
4. Combined with disturbance of consciousness;
5. Previous intracranial surgery;
6. Known or suspected cardiac dysfunction;
7. Allergic to intravenous general anesthetics;
8. Long-term history of analgesia, sedation and drug abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged between 18 and 60 years with American Society of Anesthesiology status I or II who were scheduled to receive elective surgery under general anesthesia. Patients with supratentorial glioma in right frontal lobe diagnosed by magnetic resonance imaging were included in the glioma group while patients requiring general anesthesia without intracranial-occupying lesion were included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
1. The time-frequency characteristics of EEG power changes at different sedation depths in neurosurgical patients. | Prior to anesthesia induction, three minutes after reaching the target level of sedation
  The EEG power will be calculated by raw signal at awake, eye-closed state and after reaching the steady-state sedation depths of OAA/S=3 and OAA/S=1.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing TianTan Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No